CLINICAL TRIAL: NCT04824716
Title: Evaluation of the Efficacy and Biochemical Characteristics of Ischemic Postconditioning in Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: Analysis of the Efficacy of Cardiac Ischemic Postconditioning With New Clinical End-points Using Novel Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Ferdinandy (Industry)
Collaborators: Semmelweis University Heart and Vascular Center (Other); Szeged University (Other)
Responsible Party: Sponsor-Investigator, Peter Ferdinandy, professor, Pharmahungary Group
Organization: Pharmahungary Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IPOST-01, v2.0, Nov 22, 2012
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Acute Myocardial Infarction With ST Elevation
Keywords: ischemic postconditioning; acute myocardial infarction; Investigator Initiated Trial; biomarker; coronary artery disease; ischemic; postconditioning; infarction; infarct size; area at risk; coronary occlusion; balloon catheter; percutaneous coronary intervention; PCI; MRI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease; Ischemia; Infarction; Coronary Occlusion | interventions — Ischemic Postconditioning; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postconditioning (Experimental): Patients that underwent postconditioning after primary percutaneous coronary intervention.
  Interventions: Procedure: Postconditioning
- control (Other): Patients that underwent primary percutaneous coronary intervention.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Postconditioning — The protocol of primary PCI followed by stenting is executed according to the descriptions according to the majority of relevant scientific literature on postconditioning studies and in accordance with the most recent guidelines. In the post conditioned group, after recanalization, the artery is occluded by inflation of stent balloon (4 times for 1-1 minute) followed by 1-1-minute reperfusion, repeatedly. Eight minutes after the start of examination, angiography is made in order to determine blood flow. Intervention is finished by the operator and another angiographic image is made (identical to initial standard projection).
  Arms: postconditioning
Device: Percutaneous coronary intervention — Percutaneous coronary intervention as per European Society of Cardiology guidelines.
  Arms: control

SUMMARY:
The aim of the present study was to investigate the efficacy of ischemic postconditioning in acute myocardial infarction patients. The safety of patients enrolled in the study was ensured during the entire study. Over 18 years old men and women were enrolled in the study who arrived to 2 of the most acknowledged Hungarian cardiac centres due to acute myocardial infarction and fulfilled all inclusion and exclusion criteria as per protocol. Patients in the order of their arrival were assigned either to control or post conditioned groups by turns. Medical treatment of the control group was done according to standard Percutaneous Coronary Intervention (PCI) guidelines, i.e. there was no further intervention after artery opening for 8 minutes, then stenting was performed. In the post conditioned group, after reperfusion has been confirmed, the coronary artery was occluded by inflation of the stent balloon 4 times (for 1-1 minute) followed by 1-1-minute reperfusion repeatedly to induce ischemic postconditioning. Postconditioning procedure was followed by stenting as in the control group. All other interventions and treatments in both patient groups were identical according to guidelines.

DETAILED DESCRIPTION:
Over 18 years old men and women were enrolled in the study who arrived to 2 of the most acknowledged Hungarian cardiac centres due to acute myocardial infarction and fulfilled all inclusion and exclusion criteria as per protocol. Patients in the order of their arrival were assigned either to control or post conditioned groups by turns. After closing patient enrolment, further subgrouping will be performed in case sufficient group size has been achieved as follows: (1) normal, control, (2) normal, post conditioned, (3) hypercholesterolemic, not treated with statins, control, (4) hypercholesterolemic, not treated with statins, post conditioned, (5) statin treated, control, (6) statin treated, post conditioned.

Characterisation of postconditioning is performed by the following parameters:

1. Blood tests 5 minutes before as well as 8, 60 minutes, 24 hours, and 3 months after PCI to measure nitrotyrosine, a biomarker of peroxynitrite formation (nitrosative stress) by ELISA; B-type natriuretic peptide, a biomarker of heart failure by ELISA; matrix metalloproteinase activities (MMP-2 and MMP-9) putative biomarkers of cardiac remodelling by zymography; microRNA expression pattern by sequencing and its validation by quantitative real-time polymerase chain reaction (PCR).
2. Routine laboratory tests 6, 12 and 48 hours after PCI including creatine kinase (CKMB) and cardiac troponin T (cTnT).
3. ECG immediately after recanalization and intervention after 60 and 90 minutes, then 12, 24, 36 and 48 hours later 12-lead ECG is registered.
4. Echocardiography: 48 hours after intervention, standard view to judge left ventricle segments movement disorders
5. Angiography: Blush, Syntax score, and ischemic risk zone (area at risk, AAR) are determined
6. cardiac late enhancement magnetic resonance (MR) imaging to determine infarct size

At 3-month follow-up visit the following parameters were measured: echocardiography for restitution assessment, cardiac late enhancement MR imaging to determine infarct size and cardiac function, blood sampling for above mentioned biochemical laboratory tests

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be >18 years of age
2. Myocardial infarction with elevated ST
3. Chest pain onset less than 12 hours before PCI
4. concordant ST elevation (>0,1 mV) in at least 2 ECG leads
5. Occluded main proximal or middle main coronary ('Thrombolysis In Myocardial Infarction' flow grade: 0) diagnosed with coronarography
6. Coronary opened by PCI (TIMI 2 flow grade)
7. Awake, conscious, co-operating patient, who is able to retain his breath for 10 sec
8. Signed Patient Information Leaflet and Patient Informed Consent Form

Exclusion Criteria:

1. Cardiogenic shock
2. Previous myocardial infarction in the area of the occluded coronary artery
3. Occluded coronary with visible collateral branches
4. Lack of co-operation
5. Current left or right bundle branch block (LBBB)
6. Malignant ventricle arrhythmia or atrial fibrillation
7. Killip class > 2
8. Known renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Cardiac magnetic resonance imaging | 3 months after acute myocardial infarction
  Left and right ventricular function, myocardial scar, transmurality, diffusion spectrum imaging (DSI) measurement and evaluation

SECONDARY OUTCOMES:
Echocardiography measurement of Cardiac Ejection Fraction | 48 hours and 3 months after acute myocardial infarction
  Measurement of Cardiac Ejection Fraction using Teicholz and Simpson methods on both study arms.
Echocardiography measurement of cardiac left ventricular segments for wall motion abnormalities | 48 hours and 3 months after acute myocardial infarction
  Calculation of cardiac wall motion score index on both study arms.
Laboratory measurement of blood Nitrotyrosine levels. | 5 minutes before PCI as well as 8 minutes after, 60 minutes, 6, 12, 24, 48 hours, and 3 months after acute myocardial infarction
  Laboratory measurement of Nitrotyrosine levels in blood samples with ELISA on both study arms.
Laboratory measurement of blood MMP activity. | 5 minutes before PCI as well as 8 minutes after, 60 minutes, 6, 12, 24, 48 hours, and 3 months after acute myocardial infarction
  Laboratory measurement of MMP activity in blood samples with zymography on both study arms.
Laboratory characterization of microRNA patterns with microRNA array | 5 minutes before PCI as well as 8 minutes after, 60 minutes, 6, 12, 24, 48 hours, and 3 months after acute myocardial infarction
  Laboratory characterization of microRNA expression pattern in blood samples with with microRNA array on both study arms.
Validation of selected microRNA with quantitative real-time PCR | 5 minutes before PCI as well as 8 minutes after, 60 minutes, 6, 12, 24, 48 hours, and 3 months after acute myocardial infarction
  Out of the differentially expressed microRNAs identified in Outcome 6, up to 10 different miRNAs will be selected for further validation of their specific expression change (expressed by fold-change) by quantitative real-time PCR in up to 10 randomly selected patients on both study arms, respectively.
Electrocardiography ST segment post-procedure evaluation | Post-procedure 60, 90 minutes, and 12, 24, 48 hours.
  Distortion in ST segment amplitude in millivolt (mV) and duration measured in milliseconds (ms) after procedure measured by 12-lead Electrocardiography (ECG) will be evaluated on both study arms.
Electrocardiography T wave post-procedure evaluation | Post-procedure 60, 90 minutes, and 12, 24, 48 hours.
  Distortion in T wave amplitude in millivolt (mV) and duration measured in milliseconds (ms) after procedure measured by 12-lead Electrocardiography (ECG) will be evaluated on both study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Merkely, MD, PhD, Principal Investigator — Heart and Vascular Center, Semmelweis University, Budapest; Peter Ferdinandy, MD, PhD, MBA, Study Director — Pharmahungary Group; Imre Ungi, MD, PhD, Principal Investigator — University of Szeged, Faculty of Medicine, Cardiology Center, Department of Invasive Cardiology
Locations (3):
- Hungary (3):
  - Heart and Vascular Center, Semmelweis University, Budapest
  - Pharmahungary Group, Szeged
  - Department of Invasive Cardiology of Cardiology Center, Faculty of Medicine, University of Szeged, Szeged

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of Pharmahungary Group. — http://www.pharmahungary.com
- See also: Website of Semmelweis University Heart and Vascular Center. — http://vszek.semmelweis.hu/homepage
- See also: Website of Department of Invasive Cardiology of Cardiology Center, Faculty of Medicine, University of Szeged. — http://www.med.u-szeged.hu/english